CLINICAL TRIAL: NCT02813642
Title: Evaluation of Non Traditional Cardiovascular Risk Factors in Chronic Kidney Disease Patients Starting Dialysis
Brief Title: Evaluation of Cardiovascular Risk Factors in Incident Dialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UF8851
Record Dates: First submitted 2016-06-20; First posted 2016-06-27 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease starting dialysis; cardiovascular risk; bone mineral metabolism markers
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiovascular risk evaluation (Experimental): Measurement of plasma osteoprotegerin level, plasma fibroblast growth factor 23 level, vascular calcification score and record of cardiovascular events during the 2 year follow-up
  Interventions: Biological: Plasma osteoprotegerin level; Biological: Plasma fibroblast growth factor 23 level; Procedure: Vascular calcification score

INTERVENTIONS:
Biological: Plasma osteoprotegerin level — dosage of plasma osteoprotegerin
Biological: Plasma fibroblast growth factor 23 level — dosage of plasma fibroblast growth factor 23
Procedure: Vascular calcification score — measurement of vascular calcification score by X-ray of the lateral abdominal aorta

SUMMARY:
To evaluate the relationships between bone mineral markers levels at dialysis start and vascular calcification progression during a 2 year follow up

ELIGIBILITY:
Inclusion Criteria:

* Patient who has signed the written consent form
* Patient with chronic renal failure starting dialysis therapy

Exclusion Criteria:

* Pregnancy
* Patient with chronic renal failure not yet on dialysis therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-12-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Progression of vascular calcifications during a 2 year follow up according to plasma osteoprotegerin level at inclusion | 2 years after inclusion
  osteoprotegerin will be measured in picomol/L; vascular calcifications will be measured at inclusion and after the 2 year follow up

SECONDARY OUTCOMES:
Progression of vascular calcifications during a 2 year follow up according to plasma fibroblast growth factor 23 level at inclusion | 2 years after inclusion
  fibroblast growth factor 23 will be measured in RU/milliliter; vascular calcifications will be measured at inclusion and after the 2 year follow up
Occurence of cardiovascular events during a 2 year follow up | 2 years after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Cristol, Prof, Principal Investigator — CHU Lapeyronie, Department of Biochemistry and Hormonology, Montpellier, FRANCE
Locations (5):
- France (5):
  - Centre Hémodialyse du Lez, Castelnau-le-Lez
  - AIDER, Montpellier
  - CHU Montpellier, Nephrology department, Montpellier
  - CH Nimes, Nephrology department, Nîmes
  - CH Perpignan, Nephrology department, Perpignan

IPD SHARING:
Plan to Share IPD: No